CLINICAL TRIAL: NCT00816140
Title: Comparative Study of the Levofloxacin-Based and Clarithromycin-Based Triple Therapy in First-Line Treatment for Helicobacter Pylori Eradication and Change of Gut Flora and Drug Susceptibility Before and After Treatment
Brief Title: Levofloxacin Versus Clarithromycin Triple Therapy in First-Line Treatment for Helicobacter Pylori Eradication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200702009M
Record Dates: First submitted 2007-08-06; First posted 2008-12-31 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-03

CONDITIONS: Helicobacter Infections
Keywords: Helicobacter pylori; levofloxacin; clarithromycin; ERADICATION RATE
MeSH Terms: conditions — Helicobacter Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Klaricid, triple therapy (Active Comparator): Klaricid based triple therapy
  Interventions: Drug: Klaricid based triple therapy
- Cravit, triple therapy (Experimental): Cravit based triple therapy
  Interventions: Drug: Cravit based triple therapy

INTERVENTIONS:
Drug: Cravit based triple therapy — Levofloxacin based triple therapy
  LALa regimen: levofloxacin 750mg (levofloxacin500 1.5 tablets) once daily, amoxicillin 1000mg twice daily, lansoprazole 30mg twice daily for 7 days
  Arms: Cravit, triple therapy
Drug: Klaricid based triple therapy — Clarithromycin based triple therapy
  CALa regimen: clarithromycin 500mg twice daily, amoxicillin 1000mg twice daily, and lansoprazole 30mg twice daily for 7 days
  Arms: Klaricid, triple therapy

SUMMARY:
Clarithromycin-based triple therapy containing a proton-pump inhibitor (PPI) twice daily, amoxicillin 1g twice daily, and clarithromycin 500 mg twice daily for 7 days is one of the standard firs-line therapy for Helicobacter pylori eradication. However, because of unsatisfactory eradication rate (80-85%), the Maastricht III guideline recommended extending the treatment duration to increase the eradication rate. Recently, levofloxacin (500 mg qd)-based triple therapy has been shown to achieve an eradication rate of 90% for both the first- and second-line treatment for H. pylori eradication. Several studies have demonstrated that high dose (750mg) and short-course (5 days) levofloxacin is as effective and well tolerated as traditional dose (500mg) and course (10 days) for treatment of mild-to-severe community acquired pneumonia. The high dose and short-course therapy has the potential to increase patient compliance and reduce bacterial resistance to fluoroquinolones. However, whether increasing the dosage of levofloxacin from 500mg to 750 mg qd can augment the efficacy of triple therapy in eradication of H. pylori and shorten the duration of therapy remains unknown. Although levofloxacin-based regimen was presumed to be more effective, previous reports pointed the concern that resistance to fluoroquinolone and other antibiotics which susceptible to the pumping efflux of bacteriae would increase among the gut flora.

DETAILED DESCRIPTION:
Determination of H. pylori status Prior to enrollment, the status of H. pylori infection will be determined by (1) rapid urease test (CLO test, Kimberly-Clark, USA) from antrum biopsy, (2) histological examination (Giemsa stain) of antral and body samples (two from the antral mucosa and two from the corpus mucosa), and (3) culture. Positive in any two of the three tests will be defined as positive for H. pylori infection. After-treatment H. pylori status will be determined by 13C-Urea Breath Test (13C-UBT) at 6 weeks after the completion of treatment. Successful eradication of H. pylori is defined as a negative 13C-UBT result.

Eradication Therapy Using a computer-generated number sequence, patients who meet the inclusion criteria and do not have any one of the exclusion criteria will be randomized to receive one of the following regimens: (1) CALa regimen: clarithromycin 500mg twice daily, amoxicillin 1000mg twice daily, and lansoprazole 30mg twice daily for 7 days, or (2) LALa regimen: levofloxacin 750mg (levofloxacin500 1.5 tablets) once daily, amoxicillin 1000mg twice daily, lansoprazole 30mg twice daily for 7 days (Figure 1). Adverse events will be recorded throughout the trial and during the follow-up period. Patients who do not return for 13C-UBT at 6 weeks after completion of treatment will be considered lost-to-follow-up and will be excluded from the per protocol (PP) analysis.

Rescue regimen for treatment failure after first-line regimen Patients who remained positive for H. pylori after the initial treatment as determined by the 13C-UBT will be followed by endoscopy. Biopsy will be done for H. pylori culture and antibiotic susceptibility test. All of them will then be treated with rescue regimen. The rescue regimens will be given in a cross-over manner (Figure 1). Patients who are treated with CALa regimen for 7 days as initial treatment will be treated with LALa regimen for 10 days as rescue treatment. Patients who are treated with LALa regimen for 7 days as initial treatment will be treated with CALa regimen for 10 days as rescue treatment.

Compliance and Adverse Effect Patients' compliance will be assessed by standardized interview at the end of treatment as well as by pill count in the medication boxes returned at the interview. Compliance is considered low when more than 20% of pills is found in the box. At enrollment, the patients will be informed of the common side effects from the studied antibiotics, including diarrhea, taste disturbance, nausea, bloating, loss of appetite, vomiting, abdominal pain, constipation, headache, and skin rash.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects or symptomatic patients with H. pylori infection who are aged greater than 20 years and are willing to received eradication therapy for H. pylori

Exclusion Criteria:

* Children and teenagers aged less than 20 years
* Previous eradication therapy for H. pylori
* History of gastrectomy
* Gastric malignancy, including adenocarcinoma and lymphoma
* Previous allergic reaction to antibiotics (amoxicillin, clarithromycin, levofloxacin) and prompt pump inhibitors (lansoprazole)
* Use of prompt pump inhibitors (lansoprazole) and antibiotics (amoxicillin, clarithromycin, levofloxacin) in the recent 4 weeks
* Active upper GI bleeding in the recent 1 week
* Contraindication to treatment drugs
* Pregnant or lactating women
* Severe concurrent disease or malignancy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Primary end-point of the study is to compare the eradication rate of levofloxacin-based therapy (LALa regimen for 7 days) to that achieved with the standard first line regimen (CALa regimen for 7 days). | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jawtown Lin, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Liou JM, Lin JT, Chang CY, Chen MJ, Cheng TY, Lee YC, Chen CC, Sheng WH, Wang HP, Wu MS. Levofloxacin-based and clarithromycin-based triple therapies as first-line and second-line treatments for Helicobacter pylori infection: a randomised comparative trial with crossover design. Gut. 2010 May;59(5):572-8. doi: 10.1136/gut.2009.198309. PMID 20427390